CLINICAL TRIAL: NCT05814016
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of a Single Intravenous Infusion of Danavorexton in Participants With Moderate to Severe Obstructive Sleep Apnea Undergoing General Anesthesia for Abdominal Surgery
Brief Title: A Study of Danavorexton in People With Obstructive Sleep Apnea After General Anesthesia for Abdominal Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision unrelated to patient safety.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-925-1501
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Sleep Apnea
Keywords: Drug Therapy; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — TAK-925

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose Danavorexton (Experimental): Participants will receive danavorexton intravenous (IV) infusion as high dose on Day 1 of the treatment period.
  Interventions: Drug: Danavorexton
- Low Dose Danavorexton (Experimental): Participants will receive danavorexton IV infusion as low dose on Day 1 of the treatment period.
  Interventions: Drug: Danavorexton
- Placebo (Placebo Comparator): Participants will receive a placebo-matching danavorexton IV infusion on Day 1 of the treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Danavorexton — Danavorexton IV infusion.
  Other Names: TAK-925
  Arms: High Dose Danavorexton; Low Dose Danavorexton
Drug: Placebo — Placebo matching danavorexton IV infusion.
  Arms: Placebo

SUMMARY:
The main aim is to see if danavorexton can help improve people's breathing in the recovery room after abdominal surgery.

DETAILED DESCRIPTION:
The drug being tested in this study is called danavorexton. Danavorexton is being tested in people who have moderate to severe obstructive sleep apnea undergoing general anesthesia for abdominal surgery.

The study will enroll approximately 180 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the three groups-which will remain undisclosed/unknown to the participant and study doctor during the study (unless there is an urgent medical need):

* Danavorexton high dose
* Danavorexton low dose
* Placebo All participants will receive an intravenous (IV) infusion on Day 1 of the treatment period.

This multi-center study will be conducted in approximately 20 sites in the United States. The overall time for participants to participate in the study will be up to approximately 12 months.

ELIGIBILITY:
Key Inclusion Criteria:

1. The participant has a body mass index (BMI) within the range of 18.5 to 50 kg/m^2, inclusive.
2. The participant has diagnosed or suspected moderate or severe obstructive sleep apnea (OSA) based on one of the criteria below:

   a. The participant has a snoring, tiredness, observed apnea, high blood pressure, body mass index, age, neck circumference, and gender questionnaire (STOP-Bang) score ≥5 at the screening visit. OR b. The participant has a diagnosis of moderate or severe OSA based on an in-clinic polysomnography (PSG) or home sleep test with an apnea-hypopnea index (AHI) or respiratory event index (REI) score of ≥15 and they have not had significant weight loss since their diagnostic test, in the judgment of the investigator.
3. The participant is scheduled for major abdominal surgery invading the intraperitoneal or retroperitoneal space (open or laparoscopic) that will require at least 1 inpatient overnight stay.
4. The participant is scheduled to undergo a surgery requiring general anesthesia and endotracheal intubation.
5. The participant's surgery, as planned, is anticipated to require use of IV opioids in the postanesthesia care unit (PACU).
6. The duration of the participant's surgery (i.e., incision to last stitch) is expected to be at least 2 hours and up to approximately 8 hours.
7. The participant has an American Society of Anesthesiologists (ASA) Classification of II to III.

Key Exclusion Criteria:

1. The participant has an AHI or REI score <15 based on in-clinic PSG test or at-home sleep test within 2 years before screening.
2. The participant is undergoing liver or kidney surgery.
3. The participant has a planned transfer to the intensive care unit (ICU) from the operating room.
4. For the participant, immediate (continuous positive airway pressure [CPAP]/ bilevel positive airway pressure [BiPAP]) use in the PACU is anticipated or planned.
5. The participant has undergone major surgery or donated or lost ≥1 unit of blood (approximately 500 mL) within 4 weeks before the screening visit.
6. The participant has received chemotherapy or radiation therapy within 4 weeks before administration of the study drug.
7. The participant has poorly controlled diabetes with an episode of ketoacidosis within 6 months of the screening visit.
8. The participant has a positive test result for hepatitis B surface antigen, hepatitis C virus (HCV), human immunodeficiency virus antibody/antigen at screening.
9. The participant has uncontrolled hypertension or unstable cardiovascular disease (presence of acute coronary syndrome, unstable angina, myocardial infarction <3 months, severe valvular disease, or severe structural heart disease), severe heart failure, or any condition requiring a pacemaker or defibrillator.
10. The participant has a screening electrocardiogram (ECG) with a QT interval with Fridericia correction method (QTcF) >450 milliseconds [ms] (for men) or >470 ms (for women).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Maintain Respiratory Stability for 120 Minutes in the Postanesthesia Care Unit (PACU) | Day 1
  Respiratory stability in the PACU will be considered as having been achieved if the participant can breathe without problems for 120 minutes in the PACU.

SECONDARY OUTCOMES:
Number of Episodes of Respiratory Instability per Participant Within 120 Minutes in the PACU | Day 1
  The number of episodes of respiratory instability during 120 minutes in the PACU will be assessed.
Plasma Concentration of Danavorexton at the End of Infusion (Ceoi) | Pre-dose within 1 hour before surgery and 24 hours post start of the infusion up to Day 2
Number of Participants with At Least One Occurrence of Treatment-Emergent Adverse Events (TEAEs) | Up to 12 months
  TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a study intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the study intervention or medicinal product.
Number of Participants with At Least One Occurrence of ≥1 Markedly Abnormal Value (MAV) in Post-Study Drug Laboratory Values | Up to 12 months
Number of Participants with At Least One Occurrence of ≥1 MAV in Post-Study Drug Vital Signs | Up to 12 months
Number of Participants with At Least One Occurrence of ≥1 MAV on Post-Study Drug ECGs | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (19):
- United States (19):
  - Helen Keller Hospital, Sheffield, Alabama
  - Mayo Clinic - PPDS - Hospital, Phoenix, Arizona
  - UCSD, La Jolla, California
  - Cedars Sinai Medical Hospital, West Hollywood, California
  - Mayo Clinic Jacksonville - PPDS, Jacksonville, Florida
  - University of Miami - Leonard M. Miller School of Medicine, Miami, Florida
  - Medical Research Center - Clinic/Outpatient Facility, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Rush University, Chicago, Illinois
  - University of Louisville - Hospital, Louisville, Kentucky
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Inspira Health, Mullica Hill, New Jersey
  - NYU Langone, Mineola, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Hospital, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/3861381ef14b4cde?idFilter=%5B%22TAK-925-1501%22%5D